CLINICAL TRIAL: NCT00546767
Title: Multi-Center Trial to Evaluate Home-Based Assessment Methods for Alzheimer Disease Prevention Research in People Over 75 Years Old
Brief Title: Home-Based Assessment for Alzheimer Disease Prevention
Acronym: HBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IA0123; 1RC2AG036535 (NIH); ADC-030-HBA
Record Dates: First submitted 2007-10-11; First posted 2007-10-19 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — NFKBIZ protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Mail and Live Phone (Experimental)
  Interventions: Behavioral: Mail and Live Phone
- IVR (Experimental)
  Interventions: Behavioral: Interactive Voice Response (IVR)
- Computer Kiosk (Experimental)
  Interventions: Behavioral: Home-based Computer Kiosk
- Traditional (Active Comparator)
  Interventions: Behavioral: Traditional Evaluation Instruments

INTERVENTIONS:
Behavioral: Mail and Live Phone — This group will receive assessments of all domains by mail, except for the cognitive performance assessment which will be administered via phone by a live, trained evaluator. Medication compliance will be monitored by a written medication log which will be returned by mail with the other mail-in assessments.
  Arms: Mail and Live Phone
Behavioral: Interactive Voice Response (IVR) — In this group, participants will be asked to answer questions via an automated phone system using interactive voice recognition (IVR) and key-pad response entry. Medication compliance will be monitored by the same method. A standard large-key telephone and training in the use of the interactive phone system will be provided to all participants.
  Arms: IVR
Behavioral: Home-based Computer Kiosk — Participants at entry will receive a special Kiosk-like device for collecting assessment information and will be taught to use this device. The user interface will consist of a monitor with a touch screen and a telephone handset, similar to what is often used in museum displays. Pre-recorded instructions will be delivered through the handset as well as displayed visually on the screen. Data will be collected using the handset's high-quality microphone. Daily activity assessments of timed medication use will be obtained via an automated medication tracking device.
  Arms: Computer Kiosk
Behavioral: Traditional Evaluation Instruments — Evaluation methods typically used in clinical trials
  Arms: Traditional

SUMMARY:
The purpose of this study is to evaluate three methods of performing home-based assessments in Alzheimer's Disease (AD) prevention trials. The initial in-person assessment will be done in the clinic or at home.

DETAILED DESCRIPTION:
There is an unmet need for effective, efficient, and economical methods for conducting AD prevention trials. Traditional in-person visits to clinical assessment sites are time consuming and costly and may exclude some people from participation, such as those who are older, or are less mobile or with significant medical illnesses. These may be the people who are at greatest risk for cognitive decline, and also may be without financial resources for services such as transportation to a study site. Prevention trials require long observation periods and these same issues of health, resources, and transportation may cause significant drop out. These obstacles increase expense of clinical trials which require large sample sizes, costly clinical staff and long observation periods. Thus, home-based assessments may lead to more representative recruitment of those most at risk for decline, as well as better retention and reduced study costs.

This is a randomized study of 600 participants, comparing three methods of test administration and data collection. Each enrolled participant will have an In-person (Standard) assessment (in the clinic or at home) prior to baseline.

Participants will be classified as either normal or MCI (Mild Cognitive Impairment) and randomly assigned to an assessment method and to a frequency of assessment. Cognitive performance, self-rated cognitive complaint, functioning in daily life, affective symptoms, global change, quality of life and resource use will all be assessed in each method at each visit. The total time for the at-home assessments will be approximately 45 minutes. In addition, all participants will be provided a multi-vitamin to be taken twice a day, and a measure of medication adherence will be collected for each assessment method.

Changes in certain cognitive measures may "trigger" an in-person assessment, in which participants may change from a categorization of normal or amnestic MCI, to non-amnestic MCI, impaired not MCI, or dementia (i.e., specifically Alzheimer's Disease or another dementia). We estimate that 12% of the study population will trigger over the 4 years of the study and will progress to a more impaired diagnostic category. In addition, a random sample of non-triggered cases (25%) will be selected for an in-person re-assessment during the 4 years of the protocol as a comparison for the trigger group. At the end of the 4-year study period all participants will undergo an in-person evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 and older
* Willing to sign consent
* Willing to take multi-vitamins provided by the study
* Minimal computer skills or willingness to learn (as demonstrated by completion during screening of a demonstration module for each arm)
* English fluency
* MMSE greater than 26
* Able to answer and dial a telephone
* Able to complete the in-person assessment
* Able to complete the computerized assessment including adequate speech, hearing and vision
* Independently living adults, defined as living in a setting in which the participant can ensure access to the resources for study procedures
* Participation of a study partner is desirable and encouraged, but not required

Exclusion Criteria:

* Dementia
* Use of prescription cognitive-enhancing drugs at entry (e.g. Aricept, Razadyne, Exelon, Namenda)
* Intent to continue use of own multi-vitamins (for the duration of the study participants must agree to take only study-distributed multi-vitamins)
* History or presence of major psychiatric, neurological or neurodegenerative conditions associated with significant cognitive impairment such as major stroke, Parkinson's disease, Multiple Sclerosis or Huntington's disease. Transient Ischemic Attack (TIA) is acceptable if over 6 months ago
* Medical conditions associated with life expectancy of less than 5 years
* Transient domicile interfering with ability to collect study-related data
* Current participation in a clinical trial involving Central Nervous System (CNS) medications or cognitive testing that would interfere with the current protocol (participation in Uniform Data Set (UDS) assessments by an ADC is permitted)
* Cohabitation with another participant in this particular study

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 640 (Actual)
Dates: Start 2007-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Feasibility Data -- the number of subjects recruited, screened, enrolled, and retained | 4 years
Efficiency Data -- staff time required to successfully complete data collection | Each experimental visit
Transition from cognitive health to impairment | 4 years
Method-Specific Adherence, including medication adherence | 4 years
Rate of change in domains of assessment | 4 years

SECONDARY OUTCOMES:
Research blood samples | 4 years
Safety Assessments: symptom checklist and adverse event checklist | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sano, PhD, Principal Investigator — Mount Sinai Medical School
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sun Health Reseach Institute, Sun City, Arizona
  - University of California, Irvine Institute for Brain Aging and Dementia, Irvine, California
  - University of California-San Diego ADRC/Neurosciences, La Jolla, California
  - University of California, Davis, Martinez, California
  - Stanford University / PAIRE, Palo Alto, California
  - Yale University Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville Neurology, Jacksonville, Florida
  - Wien Center, Miami Beach, Florida
  - University of South Florida, Suncoast Alzheimer's & Gerontology Center, Tampa, Florida
  - Northwestern University Cognitive Neurology & Alzheimer's Disease, Chicago, Illinois
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kentucky Sanders-Brown Center on Aging, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University Alzheimer's Disease Clinical and Research Program, Boston, Massachusetts
  - University of Michigan Psychiatry - Neuropsychology, Ann Arbor, Michigan
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - New York University Aging and Dementia Research Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Neurological Care of CNY, Syracuse, New York
  - Wake Forest University Gerontology and Geriatric Medicine, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Geriatrics, Philadelphia, Pennsylvania
  - University of Utah Center for Alzheimer's Care, Salt Lake City, Utah

REFERENCES:
- [Background] Galasko D, Bennett DA, Sano M, Marson D, Kaye J, Edland SD; Alzheimer's Disease Cooperative Study. ADCS Prevention Instrument Project: assessment of instrumental activities of daily living for community-dwelling elderly individuals in dementia prevention clinical trials. Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S152-69. doi: 10.1097/01.wad.0000213873.25053.2b. PMID 17135809
- [Background] Mundt JC, Ferber KL, Rizzo M, Greist JH. Computer-automated dementia screening using a touch-tone telephone. Arch Intern Med. 2001 Nov 12;161(20):2481-7. doi: 10.1001/archinte.161.20.2481. PMID 11700161
- [Background] Piette JD. Interactive voice response systems in the diagnosis and management of chronic disease. Am J Manag Care. 2000 Jul;6(7):817-27. PMID 11067378
- [Background] Tornatore JB, Hill E, Laboff JA, McGann ME. Self-administered screening for mild cognitive impairment: initial validation of a computerized test battery. J Neuropsychiatry Clin Neurosci. 2005 Winter;17(1):98-105. doi: 10.1176/jnp.17.1.98. PMID 15746489
- [Background] Walsh SP, Raman R, Jones KB, Aisen PS; Alzheimer's Disease Cooperative Study Group. ADCS Prevention Instrument Project: the Mail-In Cognitive Function Screening Instrument (MCFSI). Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S170-8. doi: 10.1097/01.wad.0000213879.55547.57. PMID 17135810